CLINICAL TRIAL: NCT01240460
Title: An Exploratory Pharmacodynamic Study of XL765 and XL147 Administered as Single Agents to Subjects With Recurrent Glioblastoma Who Are Candidates for Surgical Resection
Brief Title: Exploratory Study of XL765 (SAR245409) or XL147 (SAR245408) in Subjects With Recurrent Glioblastoma Who Are Candidates for Surgical Resection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TED11605; XL765-202 (Other: other study code)
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Glioblastoma; Astrocytoma, Grade IV
MeSH Terms: conditions — Glioblastoma | interventions — XL765; XL147

ARMS (3):
- 1 (Experimental): Twice-daily dosing (every 12 hours) XL765
  Interventions: Drug: XL765 (SAR245409)
- 2 (Experimental): Once-daily dosing XL147
  Interventions: Drug: XL147 (SAR245408)
- 3 (Experimental): Once-daily dosing XL765
  Interventions: Drug: XL765 (SAR245409)

INTERVENTIONS:
Drug: XL765 (SAR245409) — Supplied as 10-mg and/or 50-mg capsules
  Arms: 1; 3
Drug: XL147 (SAR245408) — Supplied as 100-mg, 150-mg and/or 200-mg tablets
  Arms: 2

SUMMARY:
The purpose of this study is to measure what effect the study drug XL765 (SAR245409) or the study drug XL147 (SAR245408) has on tumor tissue in subjects with recurrent glioblastoma (GB) who are candidates for surgical resection. XL765 (SAR245409) and XL147 (SAR245408), the two investigational agents examined in this study, XL147 (SAR245408) is a potent inhibitor of PI3 Kinase (PI3K) and XL765 (SAR245409) is a dual PI3K and mTOR inhibitor. In preclinical studies, inactivation of PI3K has been shown to inhibit growth and induce apoptosis (programmed cell death) in tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has histologically confirmed diagnosis of primary GB for which the subject has received prior treatment, including radiation and/or chemotherapy, and will be undergoing a second surgical resection.
2. The subject has available archival tumor tissue from the time of initial diagnosis of GB that is designated for central laboratory analysis.
3. The subject is ≥ 18 years old.
4. The subject has a Karnofsky performance status (KPS) ≥ 60%.
5. The subject has adequate organ and marrow function.
6. The subject has adequate fasting plasma glucose levels and glycosylated hemoglobin levels.
7. The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document.
8. Sexually active subjects (men and women) must agree to use medically-accepted barrier methods of contraception during the course of the study and for 3 months after the last dose of study drug, even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control.
9. Women of childbearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

1. The subject has confirmed secondary GB (ie, had a pathology-confirmed lower-grade glioma that subsequently recurred as a higher grade glioma).
2. The subject's tumor has a predominance of WHO Grade IV oligoastrocytoma.
3. The subject has received radiation therapy for GB within 12 weeks (≤ 84 days) before their first dose of study drug treatment.
4. The subject has received specific types of anticancer therapy (should be discussed with the treating physician)
5. The subject has not recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 Grade ≤ 1 from AEs due to surgery, radiation, antineoplastic agents, investigational drugs, or other medications that were administered before screening (except Grade 2 alopecia and Grade 2 lymphocytopenia).
6. The subject is receiving > 1 mg/day warfarin (or equivalent of other coumarin derivatives) and is unable to switch to low molecular weight heparin within 14 days before the first dose of study drug.
7. The subject is receiving enzyme-inducing anti-epileptic agents (EIAED; eg, carbamazepine, phenytoin, phenobarbital, or primidone) or valproic acid and is unable to convert to EIAED anti-seizure agents within 14 days before the first dose of study drug.
8. The subject has uncontrolled intercurrent illness including, but not limited to:

   * Ongoing or active infection
   * Hypertension (consistent blood pressure readings of > 140 mmHg systolic or > 100 mmHg diastolic) despite optimal treatment
   * Significant cardiac arrhythmias, or a recent history of serious disease, such as either symptomatic congestive heart failure or unstable angina pectoris within 3 months, or the following events within 6 months: myocardial infarction, stroke, or transient ischemic attack.
   * Inherited or acquired bleeding diathesis
9. The subject has a baseline corrected QT interval (QTc) > 460 ms.
10. The subject is unable to undergo repeated magnetic resonance imaging (MRI) scans for any reason (eg, cardiac pacemaker or ferromagnetic metal implants).
11. The subject is known to be positive for the human immunodeficiency virus (HIV). Note: HIV testing is not required for eligibility.
12. The subject has impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study treatment (eg, ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
13. The subject is pregnant or breastfeeding.
14. The subject has a previously identified allergy or hypersensitivity to components of the study treatment formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To explore the biological effect of XL765 and XL147 measured by modulation of PI3K/ mTOR pathway readouts in GB tumor tissue | Assessed between 10 and 28 days after initiation of study drug

SECONDARY OUTCOMES:
To examine the safety profile of daily oral administration of XL765 and XL147 in subjects with recurrent GB | Assessed at every visit to the study clinic for the duration of subject's treatment
To determine the levels of XL765 and XL147 in plasma and GB tumor tissue | Assessed at periodic visits between 10 and 28 days after initiation of study drug for the duration of subject's treatment
To assess the anti-proliferative and pro-apoptotic effects of XL765 and XL147 on tumor cells | Assessed at periodic visits to the study clinic for the duration of subject's treatment
To measure changes in tumor after surgery in subjects receiving XL765 and XL147 | Assessed at periodic visits following surgery 10 to 28 days after initiation of study drug for the duration of subject's treatment
To conduct genetic analyses of GB tumor tissue comparing, where feasible, tumor tissue removed during the on-study resection with tissue removed during the initial surgical resection | Assessed 10 to 28 days after initiation of study drug
To evaluate the pharmacodynamic effects of XL765 and XL147 in blood and/or blood cells for identification and characterization of surrogate biomarkers associated with the biological effects of XL765 and XL147 | Assessed at periodic visits to the study clinic
To explore the relationship between clinical response and genomic and proteomic biomarkers in the PI3K and EGFR pathways | Duration of the study (approximately 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- United States (4):
  - Investigational Site Number 840001, Los Angeles, California
  - Investigational Site Number 840003, San Francisco, California
  - Investigational Site Number 840004, Boston, Massachusetts
  - Investigational Site Number 840002, New York, New York